CLINICAL TRIAL: NCT02381028
Title: Topical Treatment With Fresh Human Milk Versus Emollient on Atopic Eczema Spots in Young Children: A Small, Randomized, Split Body, Controlled, Blinded Pilot Study
Brief Title: Topical Treatment With Fresh Human Milk Versus Emollient on Atopic Eczema Spots in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Teresa Løvold Berents, Medical doctor, Oslo University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 08/318b
Record Dates: First submitted 2015-02-28; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Atopic Eczema
Keywords: Atopic eczema; Human milk; Topical treatment; Children
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Milk, Human

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study area (Experimental): Human milk and emollient: Apobase creme® (Actavis Norway AS)
  Interventions: Other: Human milk and emollient: Apobase creme® (Actavis Norway AS); Other: Emollient: Apobase creme® (Actavis Norway AS)
- Control area (Active Comparator): Emollient: Apobase creme® (Actavis Norway AS)
  Interventions: Other: Emollient: Apobase creme® (Actavis Norway AS)

INTERVENTIONS:
Other: Human milk and emollient: Apobase creme® (Actavis Norway AS) — Topical application of human milk followed by emollient
  Arms: Study area
Other: Emollient: Apobase creme® (Actavis Norway AS) — Topical application of emollient

SUMMARY:
The aim of this small pilot study is to assess the potential effects and risks of applying fresh human milk locally on eczema spots in children with atopic eczema. This is a split body, controlled, randomized and physician blinded pilot study, of children with atopic eczema with two similar contralateral eczema spots having a mother breastfeeding the child or a sibling. Fresh expressed milk and emollient is to be applied on the intervention spot and emollient alone on the control area, three times a day for four weeks. Severity and area of the eczema spots is evaluated weekly, and samples from milk and the spots were analysed weekly with respect to bacterial colonisation.

ELIGIBILITY:
Inclusion Criteria:

* Children with atopic eczema according to Hanifin and Rajkas criteria with a mother breastfeeding the child or a sibling.
* The eczema spots in the treatment and control areas were to be similar in features and extent as well as being localized on contralateral parts of the body.

Exclusion Criteria:

* Children were excluded if the severity of the eczema spots indicated need for treatment with antibiotics and/or steroids.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Proportional change in area of the eczema spot from baseline | four weeks
  The primary outcome was proportional change in area (cm2) of the eczema spot from baseline, as measured by Visitrak™ (Smith & Nephew), a portable device used to measure the area of wounds.

SECONDARY OUTCOMES:
Transmission of bacteria from mother's milk to eczema spots in the child | four weeks
  The secondary outcome was to assess transmission of bacteria from mother's milk to eczema spots in the child.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa L Berents, MD, Principal Investigator — Oslo University Hospital

REFERENCES:
- [Derived] Berents TL, Ronnevig J, Soyland E, Gaustad P, Nylander G, Loland BF. Topical treatment with fresh human milk versus emollient on atopic eczema spots in young children: a small, randomized, split body, controlled, blinded pilot study. BMC Dermatol. 2015 May 4;15:7. doi: 10.1186/s12895-015-0027-9. PMID 25935520